CLINICAL TRIAL: NCT02080793
Title: STUDY OF PREFERENCES IN MEN FACED WITH THE DIFFERENT TREATMENT OPTIONS FOR LOCALIZED PROSTRATE CANCER WITH A GOOD OR INTERMEDIATE PROGNOSIS
Acronym: CALIPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Purpose: Other
Other Study IDs: LEJEUNE-CORMIER INCA 2012
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Patients Seen at a Urology Consultation
MeSH Terms: interventions — Surveys and Questionnaires

ARMS (2):
- Patients phase pilote (Other)
  Interventions: Other: Questionnaire
- Patients phase réelle (Other)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
This study will be based on two questionnaires

1. One specific questionnaire that has already been developed from social sciences interviews conducted in men who have been treated for localized prostrate cancer, with a good or intermediate prognosis. This questionnaire comprises 11 pairs of scenarios. Each scenario gathers in a random manner, the modalities of 7 possible characteristics of the management strategy for localized prostrate cancer, with a good or intermediate prognosis:

   * the risk of death at 5 years (modalities: 5%, 15%),
   * the risk of impotence (modalities: 0%, 25%, 50%, 75%),
   * the presence of urinary leaks (modalities: no protection during the day, one protection pad per day, several protection pads per day),
   * the duration and frequency of care provided (modalities: 2 days of care in your whole life, 7 days of care in your whole life, 5 half-days of care per week for 8 weeks, every 3 months for 2 years then every 6 months for life),
   * ablation of the prostate (modalities: Yes, No),
   * the existence of possible treatments in case of aggravation or recurrence (modalities: Yes, No),
   * the nature of the technology used (modalities: innovative technology, standard technology).

   The objective is to ask each participant of the study for each pair of scenarios, to choose from the two scenarios (binary-choice survey), the scenario he prefers.
2. The "Spielberger Inventory Trait" scale to evaluate stable characteristics in the propensity to anxiety in study participants.

ELIGIBILITY:
Inclusion Criteria:

Men:

* aged 50 to 70 years
* seen at a urology consultation
* able to understand written and spoken French
* who have provided written informed consent

Exclusion Criteria:

Men:

* under guardianship or wards of court
* who have already been diagnosed withor treated for prostrate cancer
* with recently diagnosed cancer or on treatment for this cancer

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2013-05-25 (Actual); Primary Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
Identification of personal factors linked to the management strategy chosen with regard to the preferences of patients. | Baseline

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique St Marie, Chalon-sur-Saône
  - CHU de DIJON, Dijon
  - Hôpital TENON, Paris
  - CHU de TOURS, Tours